CLINICAL TRIAL: NCT04549909
Title: Is Biochemical Pregnancy Loss Associated to Embryo or Endometrium? A Multicenter Retrospective Study
Brief Title: Biochemical Pregnancy Loss. A Multicenter Retrospective Study
Acronym: BPL
Status: Completed | Type: Observational
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); IVI Madrid (Other); Fundación IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 1902-VGO-019-EM
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy Loss, Early
Keywords: pregnancy; abortion; bioquemical
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- preimplantation genetic testing for aneuploidy (PGT-A) Group: Patients who have undergone preimplantation genetic testing for aneuploidy (PGT-A) (transfer of own frozen embryo)
  Interventions: Other: collect retrospectively data
- endometrial receptivity array (ERA) Group: Patients who have undergone frozen embryo transfer (FET) with endometrial receptivity array (ERA) test (embryos from own or donated oocytes)
  Interventions: Other: collect retrospectively data
- CONTROL OWN (CO) Group: Control group of FET from own oocytes (without ERA or PGT-A)
  Interventions: Other: collect retrospectively data
- CONTROL DONATED(CD) Group: Control group of FET from donated oocytes (without ERA or PGT-A)
  Interventions: Other: collect retrospectively data

INTERVENTIONS:
Other: collect retrospectively data — Analyse the incidence of BPL in these populations

SUMMARY:
Biochemical pregnancy loss (BPL) is a very frequent issue in human reproduction. After the implantation of the embryo, hCG disappears very soon from the maternal bloodstream and no evidence of a clinical pregnancy is seen. Different studies showed that factors such as age, oocyte and embryo quality, and endometrium receptivity may have something to do with the occurrence of biochemical pregnancy loss post assisted reproduction treatment.

The main aim of this study is to evaluate the incidence of biochemical pregnancy loss (BPL) in three different cohort populations; patients undergoing frozen embryo transfer (FET) from own oocytes after preimplantation genetic testing for aneuploidy (PGT-A), patients undergoing FET from own and donated oocytes and with endometrial receptivity array (ERA), and patients undergoing FET from own or donated oocytes (without PGTA or ERA test).

We will analyse the incidence of BPL in these populations and try to determine the role of the euploid status embryo in the first group, the endometrium in the second group and the third one as control group. We are waiting to find the value of both players in the origin of BPL.

DETAILED DESCRIPTION:
Human embryo implantation is a poorly understood process. Once the embryo implants in the endometrium, it starts to secrete hCG that can be measured in the maternal blood as early as 9 days after implantation. Only a minimal number of pregnancies get to newborn, and the majority are lost before reach the first trimester (Larsen et al., 2013).

We are looking for the role of the embryo after controlling its chromosomal ploidy, and the endometrium after controlling its transcriptomic expression. We will also use a no exposed group to the controlled euploid embryo factor neither endometrial factor that is the oocyte donation group. This analysis expects to provide more information about the key role of embryo or endometrium in BPL.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following selection criteria:

* IVF/ICSI patients aged between 18 and 44
* BMI 18-30 kg/m2
* Frozen embryo transfer from own oocytes after PGT-A
* Frozen embryo transfer with ERA test (from own or donated oocytes)
* Frozen embryo transfer (from own or donated oocytes)
* Single embryo transfer (SET) in all cycles
* Patients without uterine malformations
* Patients without recurrent miscarriage (≥ 3)
* Patients with adequate endometrial thickness (> 7mm)
* Patients without thyroid autoimmunity
* Patients without thrombophilia
* Exclude cycles with exclusively PGT-M
* Exclude FET in ovarian stimulated cycles

Exclusion Criteria:

Exclude cycles with exclusively PGT-M Exclude FET in ovarian stimulated cycles

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients who come to participating centres for assisted reproduction treatments. Patients will be divided into 4 groups according to the treatment carried out: PGT-A, ERA, FET from own oocytes (CO) or FET from donated oocytes (CD).
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Biochemical pregnancy loss (BPL) | Since 2013 to april 2019
  when the maternal serum levels of β-hCG are higher than 10 UI/L, but in the transvaginal ultrasound is not possible to appreciate any gestational structure (dichotomous qualitative variable: yes/no). This variable is considered as the fraction between patients whose β-hCG is higher than 10 UI/L, without clinically recognized pregnancy, by number of pregnant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elkin DR Muñoz, MD, Principal Investigator — IVI Vigo
Locations (1):
- IVI Vigo, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Diaz-Gimeno P, Horcajadas JA, Martinez-Conejero JA, Esteban FJ, Alama P, Pellicer A, Simon C. A genomic diagnostic tool for human endometrial receptivity based on the transcriptomic signature. Fertil Steril. 2011 Jan;95(1):50-60, 60.e1-15. doi: 10.1016/j.fertnstert.2010.04.063. Epub 2010 Jul 8. PMID 20619403
- [Derived] Munoz E, Taboas E, Alvarez M, Gil E, Perez A, Portela S, Martinez-Chapela M, Saucedo E, Garrido N. Is biochemical pregnancy loss associated with embryo or endometrium? A retrospective cohort study in frozen single embryo transfer of own and donated oocytes. Hum Reprod. 2024 May 22:deae106. doi: 10.1093/humrep/deae106. Online ahead of print. PMID 38775331